CLINICAL TRIAL: NCT01855035
Title: A Prospective, Randomised, Controlled Study to Determine the Detection of Atrial Fibrillation by Prolonged and Enhanced Holter Monitoring as Compared to Usual Care in Stroke Patients
Brief Title: Finding Atrial Fibrillation in Stroke - Evaluation of Enhanced and Prolonged Holter Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Find-AF randomised
Record Dates: First submitted 2013-05-07; First posted 2013-05-16 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Stroke
Keywords: ischemic stroke; ECG monitoring; atrial fibrillation (/flutter)
MeSH Terms: conditions — Stroke; Ischemic Stroke; Atrial Fibrillation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- prolonged ECG monitoring (Experimental): Prolonged ECG monitoring: 10-day Holter ECG at months 0, 3 and 6
  Interventions: Other: prolonged ECG monitoring
- standard care (Other): Usual care according to current guidelines (minimum of 24 hours of cardiac monitoring).
  Interventions: Other: standard care

INTERVENTIONS:
Other: prolonged ECG monitoring — 10-day Holter ECG measurement
  Arms: prolonged ECG monitoring
Other: standard care — Usual care according to current guidelines (minimum of 24 hours of cardiac monitoring).
  Arms: standard care

SUMMARY:
The purpose of this study is to assess whether repeated enhanced and prolonged ECG monitoring after ischemic stroke results in a higher detection of atrial fibrillation (/flutter) compared to usual care (at least 24 hour of cardiac monitoring).

ELIGIBILITY:
Inclusion Criteria:

* Recent cerebral ischemia defined as stroke (sudden focal neurologic deficit lasting > 24h consistent with the territory of a major cerebral artery and categorised as ischemic) and/or a corresponding lesion on brain imaging.
* Stroke symptoms started ≤ 7 days ago.
* Age ≥ 60 years.
* Modified Rankin scale ≤ 2 (prior to index event).

Exclusion Criteria:

* Known history of atrial fibrillation/flutter or atrial fibrillation/flutter on admission ECG.
* Indication for oral anticoagulation at randomisation.
* Absolute contra-indication against oral anticoagulation at randomisation.
* Intracerebral bleeding in medical history.
* Patient scheduled for Holter-ECG or cardiac Event-Recording monitoring ≥ 48 hours.
* Significant carotid artery or vertebral artery stenosis > 50% (NASCET classification), significant intracranial artery stenosis suspicious of atherosclerotic origin or acute arterial dissection explanatory of stroke symptoms.
* Implanted pacemaker device or cardioverter/defibrillator.
* Life expectancy < 1 year for reasons other than stroke (e.g. metastatic cancer).
* Concomitant participation in other controlled randomised trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2013-05; Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
number of atrial fibrillation/flutter | 30 month after study start
  The primary endpoint is the detection of newly diagnosed atrial fibrillation/flutter within 6 months and before occurrence of recurrent stroke or systemic embolism in the treatment group compared to control group.

SECONDARY OUTCOMES:
number of atrial fibrillation (/flutter) within 12 months after patient's inclusion | 24 months after study start
  Detection of newly diagnosed atrial fibrillation (/flutter) as defined for the primary endpoint but within 12 months after patient's inclusion. As patients are recruited for 12 months, this outcome measure is determined 24 months after study start.
number of atrial fibrillation (/flutter) without hospitalisation | 30 months after study start
  Detection of newly diagnosed atrial fibrillation (/flutter) as defined for the primary endpoint with the exception that hospitalisation for atrial fibrillation (/flutter) will be considered as censoring.
number of recurrent stroke or systemic embolism | 24 months after study start
  Recurrent stroke or systemic embolism within 12 months after patient's inclusion. As patients are recruited for 12 months, this outcome measure is determined 24 months after study start.
total mortality | 24 months after study start
  Total death within 12 months after patient's inclusion. As patients are recruited for 12 months, this outcome measure is determined 24 months after study start.
number of cardiovascular deaths | 24 months after study start
number of cerebrovascular deaths | 24 months after study start
number of transient ischemic attacks | 24 months after study start
number of myocardial infarctions | 24 months after study start
number of bleeding complications | 24 months after study start
quality of life | 24 months after study start
number of atrial fibrillation (/flutter) in extended monitoring period | 24 months after study start
  Incremental detection of atrial fibrillation (/flutter) in the extended Holter monitoring periods after 3 and 6 months.
costs | 24 months after study start
number of correct monitorings | 24 months after study start
  To assess the feasibility of monitoring procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Wachter, PD Dr. med., Principal Investigator — Dept. of Cardiology and Pneumology, University Medical Center Goettingen; Klaus Gröschel, PD Dr.med., Principal Investigator — Clinic and Policlinic for Neurology, University of Mainz
Locations (4):
- Germany (4):
  - Dept. of Cardiology and Pneumology, University Medical Center Goettingen, Göttingen
  - Clinic and Policlinic for Neurology, University of Mainz, Mainz
  - Dept. of Neurology, Nordwest-Hospital Sanderbusch, Sande
  - Dept. of Neurology, HSK, Dr. Horst-Schmidt-Hospital, Wiesbaden

REFERENCES:
- [Background] Wachter R, Groschel K, Gelbrich G, Hamann GF, Kermer P, Liman J, Seegers J, Wasser K, Schulte A, Jurries F, Messerschmid A, Behnke N, Groschel S, Uphaus T, Grings A, Ibis T, Klimpe S, Wagner-Heck M, Arnold M, Protsenko E, Heuschmann PU, Conen D, Weber-Kruger M; Find-AF(randomised) Investigators and Coordinators. Holter-electrocardiogram-monitoring in patients with acute ischaemic stroke (Find-AFRANDOMISED): an open-label randomised controlled trial. Lancet Neurol. 2017 Apr;16(4):282-290. doi: 10.1016/S1474-4422(17)30002-9. Epub 2017 Feb 8. PMID 28187920
- [Background] Weber-Kruger M, Gelbrich G, Stahrenberg R, Liman J, Kermer P, Hamann GF, Seegers J, Groschel K, Wachter R; Find-AF(RANDOMISED) investigators. Finding atrial fibrillation in stroke patients: Randomized evaluation of enhanced and prolonged Holter monitoring--Find-AF(RANDOMISED) --rationale and design. Am Heart J. 2014 Oct;168(4):438-445.e1. doi: 10.1016/j.ahj.2014.06.018. Epub 2014 Jul 3. PMID 25262252
- [Derived] Sadlonova M, Wasser K, Nagel J, Weber-Kruger M, Groschel S, Uphaus T, Liman J, Hamann GF, Kermer P, Groschel K, Herrmann-Lingen C, Wachter R. Health-related quality of life, anxiety and depression up to 12 months post-stroke: Influence of sex, age, stroke severity and atrial fibrillation - A longitudinal subanalysis of the Find-AFRANDOMISED trial. J Psychosom Res. 2021 Mar;142:110353. doi: 10.1016/j.jpsychores.2020.110353. Epub 2021 Jan 2. PMID 33421630
- [Derived] Wasser K, Weber-Kruger M, Groschel S, Uphaus T, Liman J, Hamann GF, Kermer P, Seegers J, Binder L, Gelbrich G, Groschel K, Wachter R. Brain Natriuretic Peptide and Discovery of Atrial Fibrillation After Stroke: A Subanalysis of the Find-AFRANDOMISED Trial. Stroke. 2020 Feb;51(2):395-401. doi: 10.1161/STROKEAHA.119.026496. Epub 2019 Dec 9. PMID 31813354
- [Derived] Wasser K, Weber-Kruger M, Jurries F, Liman J, Hamann GF, Kermer P, Uphaus T, Protsenko E, Seegers J, Mende M, Groschel K, Wachter R. The cardiac diagnostic work-up in stroke patients-A subanalysis of the Find-AFRANDOMISED trial. PLoS One. 2019 May 9;14(5):e0216530. doi: 10.1371/journal.pone.0216530. eCollection 2019. PMID 31071137

DOCUMENTS (1):
  • Study Protocol (2014-07-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT01855035/Prot_000.pdf